CLINICAL TRIAL: NCT03953625
Title: Interest of the Return to Primary Care of the "Low Back Booklet" of Health Insurance in the Recovery of Common Acute Low Back Pain
Brief Title: Interest of the Return to Primary Care of the "Low Back Pain Booklet" of Health Insurance in the Recovery of Common Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Livret lombalgie
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
Keywords: Common Acute Low Back Pain; Low Back Pain Booklet; Health Insurance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no delivery of the low back pain booklet (No Intervention): When a patient arrives at the GHPSJ emergency room or in general medical consultation at the CMT and a diagnosis of common acute low back pain is made, the physician verifies the study selection criteria.
  if the patient is included and depending on the week of inclusion, he will then be randomized to either the "no booklet" or the "booklet" group.
  If it is randomized to the arm 1 "no booklet" group, the patient will have classic management.
  All patients will be informed about the existence of the booklet. A link to the digital version on the ameli.fr website is included in the information note The patient will be contacted 3 months later by a Clinical Research Associate (CRA) to conduct a data collection.
- delivery of the low back pain booklet (Experimental): When a patient arrives at the GHPSJ emergency room or in general medical consultation at the CMT and a diagnosis of common acute low back pain is made, the physician verifies the study selection criteria.
  If the patient is included and depending on the week of inclusion, the patient will then be randomized to either the "no booklet" or the "booklet" group.
  If it is randomized in the arm 2 "with booklet" group, the management will be the same as for the "without booklet" group but with the hand delivery of the booklet in addition.
  All patients will be informed about the existence of the booklet. A link to the digital version on the ameli.fr website is included in the information note The patient will be contacted 3 months later by a Clinical Research Associate (CRA) to conduct a data collection.
  Interventions: Other: delivery of the low back pain booklet

INTERVENTIONS:
Other: delivery of the low back pain booklet — When a patient arrives at the GHPSJ emergency room or in general medical consultation at the CMT and a diagnosis of common acute low back pain is made, the physician verifies the study selection criteria.
  If it is randomized in the arm 2 "with booklet" group, the management will be the same as for the "without booklet" group but with the hand delivery of the booklet in addition.
  All patients will be informed about the existence of the booklet. A link to the digital version on the ameli.fr website is included in the information note The patient will be contacted 3 months later by a Clinical Research Associate (CRA) to conduct a data collection.
  Arms: delivery of the low back pain booklet

SUMMARY:
Low back pain is defined as pain or functional discomfort between the twelfth rib and the gluteal fold, which may be median or lateralised. It can radiate up to the thigh but never below the knee. Low back pain is said to be acute if it has been progressing for less than three months. In the acute form, it evolves on a mechanical rhythm, prevents the usual activity and occurs preferably in adults aged 20 to 55 years. 90% of these low back pains are mechanical and common, i.e. characterized by the absence of "red flags ". The red flags refer to a group of characteristic clinical signs that should alert the practitioner to the possibility of an underlying serious spinal pathology and the need for further investigation.

Common low back pain is a public health issue since it is the leading cause of health expenditure in Europe and an economic challenge (900 million euros / year and 19.1% of work stoppages in 2015 compared to 13% in 2005).

In 80% of cases, the general practitioner is in the first line of care in cases of acute low back pain. Indeed, it represents a frequent reason for consultation in general medicine (2nd reason for consultation among general practitioners in 2015).

The doctor must: track down warning signs that call into question the diagnosis of common low back pain (red flags), relieve and reassure the patient. Common low back pain very often heals spontaneously but about 10% of patients will develop chronic low back pain (persistence of pain for more than 3 months). These chronicized patients account for 80% of the total cost of low back pain.

DETAILED DESCRIPTION:
According Paracetamol is often insufficient and it is necessary to switch to level 2 analgesics (tramadol, codeine). NSAIDs are used in short courses.

It is crucial to reassure the patient about the benign nature of the condition and to insist on maintaining activities. Bed rest should never be recommended, let alone prescribed. The usual activities of daily living should be maintained as much as possible within the limits allowed by pain. A work stoppage may be considered if the professional constraints are greater than those of daily life. The return to work has no deleterious effect and must be as early as possible.

It is useful to detect early chronicization factors, especially psychosocial ones. Finally, in order to prevent lumbar disability, patient education, based on the bio-psycho-social model, must be an important part of patient care. The content of the physician's speech strongly influences the patient's beliefs and behaviour. However, if the information can be provided by the therapist, it can also be provided via brochures.

This is why the Health Insurance launched a public information campaign in November 2017 to improve the management of low back therapeutic education, pain, spine sections], the French Society of Rheumatologyk pain. The French Society of Rheumatology, The French Society of Rheumatology, therapeutic education, pain, spine sections], the French Society of Rheumatology physical and rehabilitation medicine and the college of general medicine have worked together to publish a "booklet back": I suffer from low back pain: what is it and what to do? whose main objective is to fight against false beliefs concerning inter alia "the benefits of strict rest", to promote physical activity, and to recall the true indications of complementary examinations (radiography, CT, or MRI of the spine) Thus, the back booklet intended for the patient is distributed to general practitioners via the visits of the delegates of the Health Insurance. Nearly 1,600,000 brochures were printed and made available to delegates for distribution to health professionals, with 30 brochures per general practitioner. The brochure is also available for download on ameli.fr in the "insured" and "health professionals" sections (doctors, physiotherapists, care institutions, health centres). In this study, one of the 2 participating centres is the Groupe Hospitalier Paris Saint Joseph (GHPSJ), emergency department. Also, we contacted the health insurance to receive brochures. To our knowledge, there is no other emergency service that has done this. The 2nd service centre participating in the study is the general practitioner consultation centre at the Marie-Thérèse health centre (CMT).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20 to 55 years old
* Presenting an episode of acute common low back pain diagnosed in the GHPSJ emergency room or in general medical consultation at the CMT, evolving for less than 72 hours
* Capable of giving free, informed and express consent

Exclusion Criteria:

* Existence of underlying chronic low back pain
* Associated radiculalgia descending below the knee
* Specific low back pain (with a "red flag")
* Patient not reading or understanding French
* Patient deprived of liberty
* Patient under guardianship or curatorship
* Patient under the protection of justice

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Difference in the evolution of the EIFEL score at 3 months after inclusion between the 2 patient groups | 3 months after inclusion
  A difference of 5 points in the EIFEL score between the two groups, already validated in previous studies, will be considered clinically significant.

SECONDARY OUTCOMES:
Percentage of patients who have read the booklet | 3 months after inclusion
  Differences between the 2 groups at 3 months
Percentage of patients who consulted the booklet on the ameli.fr website | 3 months after inclusion
  Differences between the 2 groups at 3 months
Percentage of patients who have resumed or started physical activity as recommended in the booklet | 3 months after inclusion
  Differences between the 2 groups at 3 months
Percentage of patients performing the recommended exercises | 3 months after inclusion
  Differences between the 2 groups at 3 months
Percentage of patients still suffering from low back pain (defined by the persistence of back pain) | 3 months after inclusion
  Differences between the 2 groups at 3 months
Numerical scale evaluating the pain | 3 months after inclusion
  Intensity of lumbar pain experienced over the last 72 hours evaluated on a numerical scale (from 0 to 10) for patients still suffering from low back pain Differences between the 2 groups at 3 months
Duration of evolution of the initial low back pain episode if resolving | 3 months after inclusion
  Differences between the 2 groups at 3 months
Duration of any work stoppage related to low back pain | 3 months after inclusion
  Differences between the 2 groups at 3 months
Number of medical consultations | 3 months after inclusion
  Differences between the 2 groups at 3 months
Number of physiotherapy or osteopathy sessions | 3 months after inclusion
  Differences between the 2 groups at 3 months
Number of additional examinations | 3 months after inclusion
  Differences between the 2 groups at 3 months
Number of analgesics taken per day during the last 72 hours (classified by WHO levels) | 3 months after inclusion
  Differences between the 2 groups at 3 months
Satisfaction with the information given about the booklet | 3 months after inclusion
  Numerical scale (from 0 to 10) Differences between the 2 groups at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: D'USSEL Marguerite, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Greenhalgh S, Selfe J. A qualitative investigation of Red Flags for serious spinal pathology. Physiotherapy. 2009 Sep;95(3):224-7. doi: 10.1016/j.physio.2009.04.006. Epub 2009 Jul 8. No abstract available. PMID 19635343
- [Result] Nicholas MK, Linton SJ, Watson PJ, Main CJ; "Decade of the Flags" Working Group. Early identification and management of psychological risk factors ("yellow flags") in patients with low back pain: a reappraisal. Phys Ther. 2011 May;91(5):737-53. doi: 10.2522/ptj.20100224. Epub 2011 Mar 30. PMID 21451099
- [Result] Bishop A, Foster NE, Thomas E, Hay EM. How does the self-reported clinical management of patients with low back pain relate to the attitudes and beliefs of health care practitioners? A survey of UK general practitioners and physiotherapists. Pain. 2008 Mar;135(1-2):187-95. doi: 10.1016/j.pain.2007.11.010. PMID 18206309
- [Result] Friedman BW, Irizarry E, Solorzano C, Khankel N, Zapata J, Zias E, Gallagher EJ. Diazepam Is No Better Than Placebo When Added to Naproxen for Acute Low Back Pain. Ann Emerg Med. 2017 Aug;70(2):169-176.e1. doi: 10.1016/j.annemergmed.2016.10.002. Epub 2017 Feb 7. PMID 28187918
- [Result] Friedman BW, Dym AA, Davitt M, Holden L, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Naproxen With Cyclobenzaprine, Oxycodone/Acetaminophen, or Placebo for Treating Acute Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 20;314(15):1572-80. doi: 10.1001/jama.2015.13043. PMID 26501533
- [Result] Coste J, Le Parc JM, Berge E, Delecoeuillerie G, Paolaggi JB. [French validation of a disability rating scale for the evaluation of low back pain (EIFEL questionnaire)]. Rev Rhum Ed Fr. 1993 May;60(5):335-41. French. PMID 8167640
- [Result] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486